CLINICAL TRIAL: NCT06460974
Title: The Effect of Stress Ball Application on Stress, Anxiety and Comfort During Chemotherapy in Women With Breast Cancer: A Randomized Controlled Study
Brief Title: The Effect of Stress Ball Application on Stress, Anxiety and Comfort During Chemotherapy in Women With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Birgul Vural Dogru, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MU-HF-BVD-02
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Patients With Breast Cancer
Keywords: Anxiety; Comfort; Breast Cancer; Stress; Stress Ball
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stress ball group (Experimental): A stress ball was applied to the patients in the stress ball group during chemotherapy treatment
  Interventions: Other: stress ball
- Control group (No Intervention): Standard care without any additional application

INTERVENTIONS:
Other: stress ball — A stress ball was applied to the patients in the during chemotherapy treatment.
  Arms: stress ball group

SUMMARY:
This research was conducted as a randomized controlled study to determine the effect of stress ball application on stress, anxiety and comfort in women with breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
The research was conducted as a randomized controlled study. A total of 74 patients were randomly assigned to the stress ball group (n=37) and the control group (n=37).

ELIGIBILITY:
Inclusion Criteria:

* who is literate in Turkish,
* who was diagnosed with stage 1, 2 and 3 breast cancer
* who had the second cure or above chemotherapy receiving treatment
* over 18 years of age
* female
* platelet level >50,000 mm3
* not having any physical problems squeezing a stress ball

Exclusion Criteria:

* those who did not agree to participate in the study
* those who received chemotherapy for the first time,
* those who had any physical disability to squeeze a stress ball
* Any receiving intravenous treatment from both arms,
* having had a unilateral or bilateral mastectomy and having a problem squeezing a stress ball,
* having any psychiatric disease,

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer | 6 months
  Distress level is determined by a visual analog scale ranging from "0-10". Patients express the psychological distress they feel with the numbers on the thermometer; "0 points" means that the patient does not experience any distress, and "10 points" means that the patient experiences the highest level of distress
State-Trait Anxiety Inventory | 6 months
  It evaluates the state of anxiety felt by the individual due to the stressful situation he is in. The first 20 items, consisting of short statements, measure the individual's state anxiety level.
General Comfort Scale | 6 months
  The scale contains a total of 48 items in a four-point Likert type and consists of four sub-dimensions (physical, psycho-spiritual, environmental, and socio-cultural sub-dimensions).

CONTACTS AND LOCATIONS:
Overall Officials: Birgül VURAL DOĞRU, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No